CLINICAL TRIAL: NCT02043782
Title: Investigation of a New 1-piece Convex Ostomy Product in Subjects With Ileostomy and Colostomy
Brief Title: Investigation of a New 1-piece Convex Ostomy Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP241
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Stoma Ileostomy; Stoma Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- First Coloplast Test (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of the treatments to the periods.
  First subjects are allocated to Coloplast Test; Secondly to either
  1. Own product (baseline)
  2. Competitor soft convex
  Interventions: Device: Coloplast Test; Device: Own product; Device: Competitor soft convex
- First Competitor soft convex (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of the treatments to the periods.
  First subjects are allocated to Competitor soft convex; Secondly to either
  1. Own product (baseline)
  2. Coloplast Test
  Interventions: Device: Coloplast Test; Device: Own product; Device: Competitor soft convex
- First Own product (Experimental): The subjects are randomised 1:1:1 into six possible treatment groups to ensure random allocation of the treatments to the periods.
  First subjects are allocated to Own product; Secondly to either
  1. Coloplast Test
  2. Competitor soft convex
  Interventions: Device: Coloplast Test; Device: Own product; Device: Competitor soft convex

INTERVENTIONS:
Device: Coloplast Test — Newly developed 1-piece convex ostomy product
Device: Own product — The subjects Own product is used as baseline performance in this investigation. The products are commercial and available on the market, and are products manufactured by manufactures who produce convex ostomy products i.e. Coloplast, Convatec, Dansac, B.Braun, Hollister and more.
Device: Competitor soft convex — A commercially available soft convex product

SUMMARY:
The aim of the investigation was to investigate the performance and safety of a new ostomy product

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age and have full legal capacity.
* Have had an ileostomy/colostomy for more than 3 months
* Have used a 1-piece flat ostomy product for the last 1 month
* Has given written Informed Consent and signed the letter of authority
* Have an ileostomy or colostomy with a diameter of 33 mm or less
* Has experienced leakage (seeping) under the baseplate at least three times during the last two weeks
* Are evaluated to be suitable for a soft convex product
* If having a colostomy: changes their product on average 2 times pr. 24h or more
* Currently uses a bag of size medi/midi or maxi

Exclusion Criteria:

* Have a loop ostomy (also called double-barrel or ostomy with two outlets).
* Are pregnant or breastfeeding
* Currently receiving or have within the past 2 month received radio- and/or chemotherapy
* Currently receiving or have within the past month received systemic or local steroid treatment in the peristomal area
* Currently suffering from peristomal skin problems (i.e. bleeding or broken skin).
* Known hypersensitivity toward any of the test products
* Participating in other interventional clinical investigations or have previously participated in this investigation
* Use irrigation during the investigation (flush the intestine with water)
* Have a fistula in the peristomal area or less than 2 cm from the edge of the baseplate
* If subject has a colostomy: empties the bag

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- TFS, Søborg, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Test - Competitor - Own: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Coloplast test product Competitor soft convex product Own product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject's own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
- Competitor - Own - Test: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Competitor soft convex product Own product Coloplast test product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject´s own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
- Own - Test - Competitor: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Own product Coloplast test product Competitor soft convex product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject´s own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
- Competitor - Test - Own: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Competitor soft convex product Coloplast test product Own product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject´s own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
- Own - Competitor - Test: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Own product Competitor soft convex product Coloplast test product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject´s own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
- Test - Own - Competitor: The subjects were randomized into six possible treatment groups:
  The order of test products for this group was:
  Coloplast test product Own product Competitor soft convex product
  Coloplast Test: Newly developed 1-piece convex ostomy product
  Own product: The subject´s own product was used as baseline performance in this investigation. The products are commercially available on the market, and are products manufactured by manufactures who produce convex ostomy products, i.e. Coloplast, Convatec, Dansac, B. Braun, Hollister and more.
  Competitor soft convex: A commercially available soft convex product
Period: Period 1
Arm/Group | Test - Competitor - Own | Competitor - Own - Test | Own - Test - Competitor | Competitor - Test - Own | Own - Competitor - Test | Test - Own - Competitor
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 6 (One subject discontinued due to an adverse event while testing own product) | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Test - Competitor - Own | Competitor - Own - Test | Own - Test - Competitor | Competitor - Test - Own | Own - Competitor - Test | Test - Own - Competitor
Started | 7 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test - Competitor - Own | Competitor - Own - Test | Own - Test - Competitor | Competitor - Test - Own | Own - Competitor - Test | Test - Own - Competitor
Started | 7 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Pooled data from all arms.
Arm/Group | All Subjects
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Region of Enrollment [Number; unit: participants]
  Denmark | 38

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is investigated on a 32-point scale (including 0 for no leakage). O represents no leakage and 32 represents the worst leakage.
Time Frame: 14 +/- 3 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Baseplates
Groups:
- Coloplast Test Product: Subjects testing Coloplast test product
- Own Product: Subjects testing own product
- Competitor Soft Convex: Subjects testing Competitor Soft Convex
Arm/Group | Coloplast Test Product | Own Product | Competitor Soft Convex
Number analyzed (Participants) | 37 | 38 | 37
Number analyzed (Baseplates) | 552 | 759 | 612
units on a scale | 2.6 (4.8) | 4.8 (5.7) | 2.5 (4.3)

ADVERSE EVENTS:
Time Frame: The AE were reported throughout the investigation, up to 5 months.
Groups:
- Coloplast Test Product: Adverse events reported by subjects testing Coloplast test product
- Own Product: Adverse events reported by subjects testing own product
- Competitor Soft Convex: Adverse events reported by subjects testing Competitor soft convex
Arm/Group | Coloplast Test Product | Own Product | Competitor Soft Convex
Serious Adverse Events (participants affected / at risk) | 1/37 | 1/38 | 0/37
Other Adverse Events (participants affected / at risk) | 22/37 | 12/38 | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=37) | Own Product (N=38) | Competitor Soft Convex (N=37)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) — Unlikely related to the product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=37) | Own Product (N=38) | Competitor Soft Convex (N=37)
Peristomal skin irritation/ broken skin/ stomal bleeding (Skin and subcutaneous tissue disorders) | 20 (26) | 5 (8) | 21 (32) — Definitely, probably or possibly related to the product
Influenza/ cold/ sore throat, Pneumonia, vomiting, infected wounds (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) — all AEs except one were unlikely or not related to the product. One AE (wound due to lower corner at hideaway scratching against leg) was definitely related to the product.
control of fistula, pain after control of fistula, constipation, sub ileus (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) — unlikely or not related to the product
headache, pain in right hand (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) — unlikely and not related to product
Herpes Zoster (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — not related to product
Cataract (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — unlikely related to product
Gash on the riight Tibia (tipped on bike) (Social circumstances) | 0 (0) | 0 (0) | 1 (1) — not related to product
(Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Its written in the AE description: drainage is something mess, due to missing flap which is on the coloplast product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes